The Presence of Ureteral Calculi Upon Supine PCNL Completion: Occlusion Balloon Catheter Versus 5FR Ureteral Catheter

PI: Mantu Gupta NCT06798753

Document Date: 12/15/2025

## 

Study ID: STUDY-24-01650 Form Version Date: 01Aug2025

**STUDY INFORMATION:** 

Study Title: The Presence of Ureteral Calculi upon supine PCNL Completion: Occlusion Balloon

Catheter versus 5FR Ureteral Catheter

Study site(s): Mount Sinai West

Lead Researcher (Principal Investigator): Mantu Gupta, MD

Physical Address: 425 W. 59th Street, Suite 4F, New York, NY 10019

Mailing Address: 425 W. 59th Street, Suite 4F, New York, NY 10019

Phone: 212-241-1272

SUMMARY OF THIS RESEARCH STUDY:

This document explains a research study you might be interested in joining. Participation in the study is voluntary. You can agree to join or not. Your decision will not limit your ability to receive care at Mount Sinai. You should only agree to take part if you understand the study and if all of your questions about the research study are answered. If you do join the study, the research team must share any new information with you that may change your mind about taking part.

The purpose of this research study is to compare the use of two different tools during kidney stone surgery (PCNL) to see which one may help reduce the presence of stone fragments in the ureter. We will look at whether using an occlusion balloon catheter (OBC) to block the exit of the kidney is helpful in preventing fragments from moving into the ureter during the procedure.

If you choose to take part, you will be randomly assigned to one of two groups. In one group, a small tube called an occlusion balloon catheter (OBC) will be inserted into your ureter at the beginning of the surgery. The OBC has a small balloon that can be inflated to help prevent stone fragments from moving into your ureter. In the other group, a 5FR ureteral catheter (5FR-UC), a small, open-ended tube, will be used to assist with the procedure. Both catheters are used as part of the standard of care for your procedure and are typically chosen based on your surgeon's preference. The rest of your surgery will follow the standard care practices. After the procedure, a flexible scope will be used to check for any stone fragments in your ureter, and if there are, they will be removed. There are no additional visits required, and your participation will end once your surgery is over. There are no costs to participating in this study, and you will not be paid to participate in this study.

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 


If you choose to take part, the main risk to you is the slight increase in surgery time and time under anesthesia due to the time it takes to check for and remove any stone fragments after the procedure. This is expected to be 5-10 additional minutes at most. There is also the risk of loss of private information, but there are procedures in place to minimize this risk.

You will not benefit directly from taking part in this research.

Instead of taking part in this research, you may have your kidney stone removal surgery without participating in the research study.

If you are interested in learning more about this study, please continue to read below.

#### STUDY PARTICIPATION:

You may qualify to take part in this research study because you are scheduled to undergo kidney stone removal surgery in the supine position.

Your participation in this research study is expected to last one day (the day of surgery).

There are 110 people expected to take part in this research study at Mount Sinai West.

Funds for conducting this research study are provided by Mount Sinai.

#### **DESCRIPTION OF WHAT IS INVOLVED:**

If you agree to take part in this research study, here is what may be involved:

- During your initial consultation with your urologist at Mount Sinai, you will be asked to read this informed consent form. The research team will also ask for permission to collect data from your medical records related to this procedure. You will have time to ask any questions about the study to your study doctor. After all your questions have been answered and you fully understand the information in the consent form, you may choose to participate by signing and dating the form.
- o On the day of surgery, you will be randomly assigned to one of two groups: OBC or 5FR-UC.
- At the start of the procedure, either the OBC or 5FR-UC will be inserted into your ureter. The rest
  of the surgery will proceed as planned, following the standard of care.
- Both the OBC and 5FR-UC are commonly used in PCNL procedures and are typically chosen based on the surgeon's preference.
- After the surgery, an additional procedure called antegrade flexible ureteroscopy will be performed to check for and remove any stone fragments from your ureter. This is an accepted and commonly

Rev 11.11.2022 (Amendment 1-03.09.2023)



## ****


used procedure during PCNL, but it is not performed in every case as part of routine care. In this study, it will be performed for all participants to ensure consistency and to assess stone clearance as part of the research study.

- No changes to your anesthesia will be made for research purposes, but you may be under anesthesia for an additional 5-10 minutes due to the time needed to check for and collect any stone fragments.
- o Once the surgery is complete, your participation in the study will also be complete.

#### Randomization

No one, not you, or anyone from your medical team or from the research team will be able to choose what ureteral catheter you get. It will be by chance, like flipping a coin. You will have an equal chance of being given either the OBC or 5FR-UC.

### **USE OF YOUR DATA AND/OR SAMPLES:**

The research team will never use or share your personal information (such as, name, address, date of birth, social security number), study data and/or samples (blood, tissue, urine, saliva, or any other body matter) that are collected as part of this study for future research, even if your identity is removed. Your data and/or samples will only be used to complete this study and then they will be destroyed.

#### YOUR RESPONSIBILITIES IF YOU TAKE PART IN THIS RESEARCH:

If you decide to take part in this research study, you will be responsible for the following things:

- Follow the directions of your doctor
- Allow the research team to access your medical records

| COSTS OR PAYMENTS THAT MAY RESULT FROM PARTICIPATION: |
|---|
| You will not be paid for taking part in this study. Being in this study will not cost you anything extra. |
| POSSIBLE BENEFITS: |
| FOR IRB USE ONLY |
| ev 11.11.2022 (Amendment 1-03.09.2023) |



## 


This study is not designed to benefit you personally. However, possible future benefits to others include helping researchers learn more about ways to optimize kidney stone removal surgery.

#### POSSIBLE RISKS AND DISCOMFORTS:

- There is a risk of increased procedure duration due to the time needed for the antegrade flexible ureteroscopy to check for and remove any stone fragments. This is expected to be 5-10 additional minutes.
- There is the risk of anesthesia exposure due to increased procedure time. The slight
  extension of the procedure time means you may be under anesthesia for an additional 510 minutes. This can increase the risk of anesthesia-related complications such as
  respiratory or cardiovascular complications, nausea, and delayed recovery. This risk is
  expected to be minimal.
- Risk of loss of private information; this risk always exists, but there are procedures in place to minimize the risk.
  - o Group Risks Although your name will not be given to researchers, basic information such as your race, ethnic group, and sex may be shared. This information helps researchers learn whether the factors that lead to health problems are the same in different groups of people. It is possible that such findings could one day help people of the same race, ethnic group, or sex as you. However, they could also be used to support harmful stereotypes or discrimination.
  - O Privacy Risks Your name and other information that could directly identify you (such as an address, date of birth, or social security number) will never be placed into a database. However, because your genetic information is unique to you, there is a small chance that someone could trace it back to you. The risk of this happening is very small, but may grow in the future. Since the database contains genetic information, a break in security may also pose a potential risk to blood relatives as well as yourself. For example, it could be used to make it harder for you (or a relative) to get or keep a job or insurance. If your private information was misused, it is possible you would experience other harms, such as stress, anxiety, stigmatization, or embarrassment from revealing information about your family relationships, ethnic heritage, or health conditions.

### OTHER OPTIONS TO CONSIDER:

You may decide not to take part in this research study. If you decide not to take part, this will not affect the clinical care you receive at Mount Sinai. The choice is totally up to you.

*Instead* of being in this research study you may have your kidney stone removal surgery without allowing the research team to randomize which ureteral catheter is used during the procedure.

------FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)




#### IN CASE OF INJURY DURING THIS RESEARCH STUDY

If you believe that being in this research study has harmed you, you should contact the Lead Researcher. Their contact information is listed at the beginning of this consent form.

#### ENDING PARTICIPATION IN THE RESEARCH STUDY:

You may stop taking part in this study at any time. No matter what you choose, your care and benefits through Mount Sinai will not be negatively impacted.

If you decide to stop being in the study, please contact the Lead Researcher or the research staff.

You may also withdraw your permission for the researchers to use and share any of your protected information for research, but <u>you must do so in writing</u> to the Lead Researcher at the address on the first page. Even if you withdraw your permission, the Lead Researcher may still use the information that was already collected if that information is necessary to complete the research study. Your health information may still be used or shared after you withdraw your authorization if you have an adverse event (a bad effect) from taking part in the research study.

If you decide you don't want your data and/or samples to be used for research anymore, you can contact the researcher and ask to have your data and/or samples withdrawn or labeled so that they will not to be used in additional projects or shared. If your data and/or samples have already been shared with researchers, those researchers will be asked to stop using them. However, if any data and/or samples have already been shared without your identity or a linking code, it won't be possible to retrieve them. Data and/or samples that have already been used will not be affected by your decision. If your data and/or samples have already been deposited in an external repository, the study team will request that your data and/or samples be removed.

<u>Withdrawal without your consent</u>: The Lead Researcher, the funder or Mount Sinai may stop your involvement in this research study at any time without your consent. This may be because the research study is being stopped, the instructions of the research team have not been followed, the Lead Researcher believes it is in your best interest, or for any other reason. If data and/or samples have been stored as part of the research study, they too can be destroyed without your consent.

| C | $\mathbf{O}$ | JT | $\Delta CT$ | INF | :ORI | МΔТ | TION: |
|---|---|---|---|---|---|---|---|
| J | VI. | <b>7</b> / | マンコ | 11.41 | $\sim$ 1 $^{\circ}$ 1 | | |

-----FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 


If you have any questions, concerns or complaints at any time about this research, or you think the research has harmed you, please contact the office of the research team and/or the Lead Researcher at phone number 212-241-1272.

#### **DISCLOSURE OF FINANCIAL INTERESTS:**

Researchers sometimes get paid for consulting or doing work for companies that produce drugs, biologics or medical devices. If you have questions regarding industry relationships, you are encouraged to talk to the Lead Researcher or visit our website at http://icahn.mssm.edu/ where Mount Sinai publicly discloses the industry relationships of our faculty.

#### MAINTAINING CONFIDENTIALITY - HIPAA AUTHORIZATION:

As part of this study, some of your private and/or protected health information will be obtained, used, and shared with your permission. There is a Federal Health Insurance Portability and Accountability Act (HIPAA) that makes sure this is done correctly and safely.

#### What is protected health information (PHI)?

PHI is the combination of two things:

- 1. PHI contains information that identifies you. It will be used to contact you and link you to your health information, like name, date of birth, medical record number, and address.
- 2. PHI also contains health information, including information about your mental and physical health from your visits to doctors or hospitals, or from study visits.

Every time you visit a hospital or your doctor, PHI is created and recorded in your medical record by your healthcare providers. In the same way, the PHI created as part of this study will be linked to who you are and your medical information.

What PHI is collected and used in this research study, and might also be shared with others?

As part of this study, the research team at the hospital(s) involved in the research will collect your, name, telephone/fax numbers, dates directly related to the individual (birth, admission, discharge, date of death, etc.), and medical records number.

During the study, the researchers will gather information by:

- Reviewing and/or taking your medical history (includes current and past medications or therapies, illnesses, conditions or symptoms, family medical history, allergies, etc.)
- Doing a physical examination that generally also includes blood pressure reading, heart rate, breathing rate, and temperature.

-----FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 


 Completing the tests, procedures, questionnaires and interviews explained in the description section of this consent.

#### Why is your PHI being used?

Researchers need the information that identifies you so they can contact you during the study. They need your health information and the results of any tests and procedures being collected as part of this study to answer the questions posed in the study. The purpose of the study is discussed earlier in this consent form. Before researchers analyze the data, they remove any information that would let others know who you are or that you took part in the study. If researchers publish or present study results at scientific meetings, lectures, or other events, their presentations would not include any information that would let others know who you are, unless you give separate permission to do so.

The Lead Researcher may also use and share the results of these tests and procedures with other healthcare providers at Mount Sinai who are involved in your care or treatment. The research team and other authorized members of The Mount Sinai Health System ("Mount Sinai") workforce may use and share your information to ensure that the research meets legal, institutional or accreditation requirements. For example:

- The Mount Sinai Program for the Protection of Human Subjects is responsible for overseeing research on human participants and may need to see your information.
- If you receive any payments for taking part in this study, the Mount Sinai Finance Department may need your name, address, social security number, payment amount, and related information for tax reporting purposes.
- If the research team uncovers abuse, neglect, or reportable diseases, this information may be disclosed to appropriate authorities.

### Who, outside Mount Sinai, might receive your PHI?

As part of the study, the Lead Researcher, research team and others in the Mount Sinai workforce may disclose your PHI, including the results of the research study tests and procedures, to the following people or organizations: (It is possible that there may be changes to the list during this research study; you may request an up-to-date list at any time by contacting the Lead Researcher.)

- The United States Department of Health and Human Services (DHHS) and the Office of Human Research Protection (OHRP) (the government organization that is responsible for protecting human research participants).

In all disclosures outside of Mount Sinai, you will not be identified by name, social security number, address, telephone number, or any other direct personal identifier unless disclosure of the direct identifier is required by law. Some records and information disclosed may be identified with a unique code number. The Lead Researcher will ensure that the key to the code will be kept in a locked file, or will be securely stored electronically. The code will not be used to link the information back to you without your permission, unless the law requires it, or rarely if the Institutional Review Board (IRB)

------FOR IRB USE ONLY-------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 


allows it after determining that there would be minimal risk to your privacy. It is possible that a sponsor or their representatives, a data coordinating office, a contract research organization, may come to inspect your records. Even if those records are identifiable when inspected, the information leaving the institution will be stripped of direct identifiers. Additionally, when applicable, the monitors, auditors, the IRB, OHRP, as well as the Food and Drug Administration (FDA) will be granted direct access to your medical records for verification of the research procedures and data. OHRP and FDA are authorized to remove information with identifiers if necessary to complete their task. By signing this document you are authorizing this access. The results of this research may be published. However, your name and other identifying information will be kept confidential.

## For how long will Mount Sinai be able to use or disclose your PHI?

Your authorization for use of your PHI for this specific study does not expire.

### Will you be able to access your records?

During your participation in this study, you will have access to your medical record and any study information that is part of that record. The research team is not required to release research information to you that is not part of your medical record.

## Do you need to give the researchers permission to obtain, use or share your PHI?

NO! If you decide not to let the research team obtain, use or share your PHI, you should not sign this form, and you will not be allowed to volunteer in the research study. If you do not sign, it will not affect your treatment, payment, or enrollment in any health plans or affect your eligibility for benefits.

### Can you change your mind?

If you decide to stop being in the study, please contact the Lead Researcher or the research staff. The research team may ask you whether they can continue to collect information from your medical record. You will also have to decide if you wish to limit the continued use of the information collected during the study. Under US privacy laws you may also withdraw your permission for the researchers to use and share any of your protected information for research, but you must do so in writing to the Lead Researcher at the address on the first page.

Even if you withdraw your permission, the Lead Researcher may still use the information that was already collected, but only to complete this research study. Your health information may still be used or shared after you withdraw your authorization if you have an adverse event (a bad effect) from taking part in the research study.

It is important for you to understand that once information is disclosed to others outside Mount Sinai, the information may be re-disclosed and will no longer be covered by the federal privacy protection regulations. However, where possible, Mount Sinai has entered into agreements with those who will receive your information to continue to protect your confidentiality.

------FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



# 


If researchers are reviewing your medical records or asking questions about your medical history or conditions, it is possible that they may learn information related to your HIV status. If that is the case, the following information concerns you. If researchers are not reviewing your medical records or asking questions about your medical history or conditions, then you may ignore the following section.

### **Notice Concerning HIV-Related Information**

If you are authorizing the release of HIV-related information, you should be aware that the recipient(s) is (are) prohibited from re-disclosing any HIV-related information without your authorization unless permitted to do so under federal or state law. You also have a right to request a list of people who may receive or use your HIV-related information without authorization. If you experience discrimination because of the release or disclosure of HIV-related information, you may contact the New York State Division of Human Rights at (888) 392-3644 or the New York City Commission on Human Rights at (212) 416-0197. These agencies are responsible for protecting your rights.

## How the Institutional Review Board (IRB) can help you:

This research has been reviewed and approved by an Institutional Review Board (IRB). You may reach a representative of the Mount Sinai Program for Protection of Human Subjects at telephone number (212) 824-8200 during regular work hours (Monday-Friday, 9am-5pm, excluding holidays) for any of the reasons listed below. This office will direct your call to the right person within the Mount Sinai Health System:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You are not comfortable talking to the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

------FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



# 


| | your permission to take part in this health information. A signed and dat | | |
|---|---|---|---|
| Signature of Participant | Printed Name of Participant | Date | Time |
| PERSON EXPLAINING STUDY | AND OBTAINING CONSENT: | | |
| Signature of Consent Delegate | Printed Name of Consent Deleg | ate Date | Time |
| | nat the information in the consent do<br>ined to, and apparently understood l<br>participant. | | |
| Signature of Witness | Printed Name of Witness | Date | Time |
| Rev 11.11.2022 (Amendment 1-03.09.20 | FOR IRB USE ONLY | | |

